CLINICAL TRIAL: NCT02017340
Title: A European Multicentre Double-blind Placebo-controlled Phase III Trial of Nilvadipine in Mild to Moderate Alzheimer's Disease
Brief Title: A Phase III Trial of Nilvadipine to Treat Alzheimer's Disease
Acronym: NILVAD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Prof Brian Lawlor (Other)
Collaborators: University of Dublin, Trinity College (Other); Molecular Medicine Ireland LBG (Unknown); Alzheimer Europe (Other); Archer Pharmaceuticals, Inc. (Industry); E-Search Limited (Unknown); University College Dublin (Other); King's College London (Other); Istituto Di Ricerche Farmacologiche Mario Negri (Other); University Hospital, Lille (Other); University of Ulm (Other); Szeged University (Other); Göteborg University (Other); University College Cork (Other); Aristotle University Of Thessaloniki (Other); Stichting Katholieke Universiteit (Other)
Responsible Party: Sponsor-Investigator, Prof Brian Lawlor, Project Coordinator, St. James's Hospital, Ireland
Organization: St. James's Hospital, Ireland (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NILVAD2012; 2012-002764-27 (EudraCT Number); 279093 (Other Grant/Funding Number: European Commission Framework Programme)
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-03

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; Investigator-driven clinical trial; Nilvadipine; Calcium Channel blocker; Elderly; Therapeutic Intervention
MeSH Terms: conditions — Alzheimer Disease | interventions — nilvadipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 250 patients will receive the placebo
  Interventions: Drug: Placebo
- Nilvadipine (Active Comparator): 250 patient will receive the active drug Nilvadipine 8mg
  Interventions: Drug: Nilvadipine

INTERVENTIONS:
Drug: Nilvadipine — 8mg of Nilvadipine taken once a day at lunch time for 78 weeks
  Other Names: Also known as Nilvadil (Brand Name)
  Arms: Nilvadipine
Drug: Placebo — 8mg Placebo tablet taken once a day at lunch time for 78 weeks
  Arms: Placebo

SUMMARY:
Alzheimer's disease (AD) is an ever-increasing public health concern among the aging population and is the most common form of dementia affecting more than 15 million individuals worldwide and around 5 million Europeans. The direct and indirect costs of AD and other dementias amount to more than €440,000 million each year (www.alz.org, 2010).

Even modest therapeutic advances that delay disease onset and progression could significantly reduce the global burden of the disease and the level of care required by patients. While there are symptomatic-based drug therapies available for AD, these medications do not prevent the disease process itself. There is therefore an imperative to develop new treatments for AD that have disease modifying effects. This double-blind placebo controlled study will test the efficacy and safety of nilvadipine in 500 subjects with mild to moderate AD over a treatment period of 18 months. There is a strong scientific rationale for this study: Nilvadipine, a licensed calcium channel enhances Aß clearance from brain and restores cortical perfusion in mouse models of AD. Nilvadipine is safe and well tolerated in AD patients and clinical studies with this medication have shown stabilization of cognitive decline and reduced incidence of AD, pointing to both symptomatic and disease modifying benefits. Male and female patients with mild to moderate AD aged between 50 and 90 with a range of medical morbidities and frailty will be included in the study. If this trial is successful, nilvadipine would represent an advance in the treatment of AD patients and would have a major impact on the health and social care costs incurred in Europe by this neurodegenerative disorder. Furthermore, the creation of the NILVAD network will support future clinical trials and research innovation in AD across Europe.

DETAILED DESCRIPTION:
Please see 'Brief Summary', above

ELIGIBILITY:
Inclusion Criteria:

1. Age range: Adult subjects, males and females over age 50 years.
2. Prior diagnosis of mild to moderate probable AD based on NINCDS-ADRDA criteria (see Appendix B) and
3. Standardised Mini-Mental State Examination (SMMSE) score > 12 on stable dose (>3 months of cholinesterase inhibitor and or memantine). Subjects who are not on cholinesterase inhibitors or memantine due to poor tolerability and/or who will not require treatment with these medications during the course of the study can be included.
4. Collateral informants such as a spouse, family member, close friend. The informant must have close contact with the subject and agree to monitor/manage study drug adherence, observe for possible adverse events, assist with psychometric measures requiring informant information, and accompany the subject to all evaluation visits.
5. Fluency in relevant language sufficient to reliably complete all study assessments.
6. Systolic BP > 100 mmHg but ≤ 159 mmHg, and diastolic BP > 65 mmHg but ≤ 99 mmHg on resting office based BP measurements, or a Systolic BP > 105 mmHg but ≤ 140 mmHg, and diastolic BP > 70 mmHg but ≤ 90 mmHg on ABPM measurement

Exclusion Criteria:

1. Subjects with co-morbid dementia due to other neurological disorders such as Parkinson's disease, vascular dementia, Huntington's disease, Pick's disease, Creutzfeldt-Jakob disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, or multiple sclerosis, as well as subjects with HIV disease, neurosyphilis, history of significant head trauma with loss of consciousness followed by persistent neurological deficits, known structural brain abnormalities, or any other condition known to interfere with cognitive function.
2. Subjects currently taking any calcium channel blocker or Beta-blocker
3. Subjects who in the opinion of the investigator, have a medical condition that would preclude them from participating in the study (e.g.hemodynamically significant coronary artery disease., chronic heart failure, syncope within the past year, significant valvular heart disease i.e. severe aortic and mitral stenosis.. symptomatic orthostatic hypotension within the last year, subjects requiring more than one agent to control BP.), or subjects who in the opinion of the investigator are unlikely to complete per protocol due to care issues etc:
4. Current Axis I diagnosis of schizophrenia, bipolar disorder, major depression. Subjects who are currently or who have within the past year met criteria for drug or alcohol abuse or dependence.
5. Pregnant women or women who may possibly become pregnant.
6. Subjects with a history of hypersensitivity to nilvadipine (Nivadil).
7. Subjects who have taken an investigational or other unapproved drug during the 30 days or five half-lives, whichever is longer, prior to baseline.
8. Subjects who are participating in other research studies.
9. Patients with a SBP of ≤ 100 mmHg and/or a DBP of ≤ 65 mmHg on office based BP measurements, or a SBP ≤ 105 mmHg and/or a DBP of ≤ 70 mmHg on ABPM will not be included in the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2013-04-24 (Actual); Primary Completion 2016-12-16 (Actual); Study Completion 2016-12-16 (Actual)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale (ADAS) Cog | 18 months
  The Alzheimer's Disease Assessment Scale (Cognitive) (Mohs et al. 1983) ADAS-cog 12 is a primary efficacy outcome measure, and includes 12 items of cognitive evaluation, namely immediate word recall, naming objects and fingers, commands, constructional praxis, ideational praxis, orientation, word recognition, remembering test instructions, spoken language ability, word-finding difficulty in spontaneous speech, comprehension & delayed recall. A higher ADAS-cog score indicates a poorer cognitive function.

SECONDARY OUTCOMES:
Clinical Dementia Rating Scale Sum of Boxes (CDR-sb) | 18 months
  Clinical Dementia Rating Scale Sum of Boxes (CDR-sb) (Morris et al 1993) is the secondary efficacy outcome measure. This is a semi-structured interview with the caregiver and the patient. The patient's performance in the domains of memory, orientation, judgment, problem solving, community affairs, home and hobbies and personal care are assessed. The CDR-sb is scored from 0-18, with the higher score indicated greater impairment.
Disability Assessment for Dementia (DAD) | 18 months
  Disability Assessment for Dementia (DAD) (Gelinas et al. 1999) is a key secondary efficacy outcome measure and evaluates the basic and instrumental activities in daily activities of elderly people with dementia. This 40-item scale addresses a range of functional domains: eating, meal preparation, telephoning, hygienic, dressing, medication, corresponding, finance, leisure, and housework.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Lawlor, Prof, Principal Investigator — University of Dublin, Trinity College
Locations (23):
- France (7):
  - Centre Hospitalier Universitaire d'Amiens (CHU Amiens), Amiens
  - Centre Hospitalier Universitaire de Bethune (CH Bethune), Béthune
  - Centre Hospitalier Universitaire de Caen (CHU Caen), Caen
  - Centre Hospitalier Universitaire de Calais (CHU Calais), Calais
  - Centre Hospitalier Universitaire de Lens (CHU Lens), Lens
  - Centre Hospitalier Regional et Universitaire de Lille (CHRU Lille), Lille
  - Centre Hospitalier Universitaire de Saint Philibert (GHICL), Lille
- University of Ulm, Ulm, Germany
- Greece (3):
  - "G. Papanicolaou" Hospital, Athens
  - "G.Papageorgiou" Hospital, Athens
  - AXEPA Hospital, Athens
- Szeged University, Szeged, Hungary
- Ireland (2):
  - University College Cork, Cork
  - St James Hospital, Dublin
- Italy (4):
  - Hospital of Brescia, Brescia
  - Hospital Castellanza, Castellanza
  - Hospital of Genoa, Genoa
  - Hospital of Milan, Milan
- Netherlands (3):
  - Hospital of Arnhem, Arnhem
  - Hospital of Maastricht, Maastricht
  - Hospital of Nijmegen, Nijmegen
- Gothenburg Univeristy, Gothenburg, Sweden
- Kings College London, London, United Kingdom

REFERENCES:
- [Background] Brogden RN, McTavish D. Nilvadipine. A review of its pharmacodynamic and pharmacokinetic properties, therapeutic use in hypertension and potential in cerebrovascular disease and angina. Drugs Aging. 1995 Feb;6(2):150-71. doi: 10.2165/00002512-199506020-00007. PMID 7711361
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Facchinetti F, Fasolato C, Del Giudice E, Burgo A, Furegato S, Fusco M, Basso E, Seraglia R, D'Arrigo A, Leon A. Nimodipine selectively stimulates beta-amyloid 1-42 secretion by a mechanism independent of calcium influx blockage. Neurobiol Aging. 2006 Feb;27(2):218-27. doi: 10.1016/j.neurobiolaging.2005.02.006. PMID 16399208
- [Background] Fleckenstein A. Specific pharmacology of calcium in myocardium, cardiac pacemakers, and vascular smooth muscle. Annu Rev Pharmacol Toxicol. 1977;17:149-66. doi: 10.1146/annurev.pa.17.040177.001053. No abstract available. PMID 326161
- [Background] Forette F, Seux ML, Staessen JA, Thijs L, Birkenhager WH, Babarskiene MR, Babeanu S, Bossini A, Gil-Extremera B, Girerd X, Laks T, Lilov E, Moisseyev V, Tuomilehto J, Vanhanen H, Webster J, Yodfat Y, Fagard R. Prevention of dementia in randomised double-blind placebo-controlled Systolic Hypertension in Europe (Syst-Eur) trial. Lancet. 1998 Oct 24;352(9137):1347-51. doi: 10.1016/s0140-6736(98)03086-4. PMID 9802273
- [Background] Forette F, Seux ML, Staessen JA, Thijs L, Babarskiene MR, Babeanu S, Bossini A, Fagard R, Gil-Extremera B, Laks T, Kobalava Z, Sarti C, Tuomilehto J, Vanhanen H, Webster J, Yodfat Y, Birkenhager WH; Systolic Hypertension in Europe Investigators. The prevention of dementia with antihypertensive treatment: new evidence from the Systolic Hypertension in Europe (Syst-Eur) study. Arch Intern Med. 2002 Oct 14;162(18):2046-52. doi: 10.1001/archinte.162.18.2046. PMID 12374512
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Furuichi Y, Takakura S, Satoh H, Mori J, Kohsaka M. The effect of nilvadipine, a dihydropyridine type calcium channel blocker, on local cerebral blood flow in rats. Jpn J Pharmacol. 1992 Apr;58(4):457-60. doi: 10.1254/jjp.58.457. PMID 1405041
- [Background] Gelinas I, Gauthier L, McIntyre M, Gauthier S. Development of a functional measure for persons with Alzheimer's disease: the disability assessment for dementia. Am J Occup Ther. 1999 Sep-Oct;53(5):471-81. doi: 10.5014/ajot.53.5.471. PMID 10500855
- [Background] Hanyu H, Hirao K, Shimizu S, Sato T, Kiuchi A, Iwamoto T. Nilvadipine prevents cognitive decline of patients with mild cognitive impairment. Int J Geriatr Psychiatry. 2007 Dec;22(12):1264-6. doi: 10.1002/gps.1851. No abstract available. PMID 18033677
- [Background] Inouye M, Mio T, Sumino K. Nilvadipine protects low-density lipoprotein cholesterol from in vivo oxidation in hypertensive patients with risk factors for atherosclerosis. Eur J Clin Pharmacol. 2000 Apr;56(1):35-41. doi: 10.1007/s002280050717. PMID 10853875
- [Background] Khachaturian AS, Zandi PP, Lyketsos CG, Hayden KM, Skoog I, Norton MC, Tschanz JT, Mayer LS, Welsh-Bohmer KA, Breitner JC. Antihypertensive medication use and incident Alzheimer disease: the Cache County Study. Arch Neurol. 2006 May;63(5):686-92. doi: 10.1001/archneur.63.5.noc60013. Epub 2006 Mar 13. PMID 16533956
- [Background] Kagawa H, Nomura S, Ozaki Y, Nagahama M, Fukuhara S. Effects of nilvadipine on cytokine-levels and soluble factors in collagen disease complicated with essential hypertension. Clin Exp Hypertens. 1999 Oct;21(7):1177-88. doi: 10.3109/10641969909052196. PMID 10513835
- [Background] Lopez-Arrieta JM, Birks J. Nimodipine for primary degenerative, mixed and vascular dementia. Cochrane Database Syst Rev. 2002;(3):CD000147. doi: 10.1002/14651858.CD000147. PMID 12137606
- [Background] Lubben J, Blozik E, Gillmann G, Iliffe S, von Renteln Kruse W, Beck JC, Stuck AE. Performance of an abbreviated version of the Lubben Social Network Scale among three European community-dwelling older adult populations. Gerontologist. 2006 Aug;46(4):503-13. doi: 10.1093/geront/46.4.503. PMID 16921004
- [Background] Maxwell CJ, Hogan DB, Ebly EM. Calcium-channel blockers and cognitive function in elderly people: results from the Canadian Study of Health and Aging. CMAJ. 1999 Sep 7;161(5):501-6. PMID 10497605
- [Background] McKhann G, Drachman D, Folstein M, Katzman R, Price D, Stadlan EM. Clinical diagnosis of Alzheimer's disease: report of the NINCDS-ADRDA Work Group under the auspices of Department of Health and Human Services Task Force on Alzheimer's Disease. Neurology. 1984 Jul;34(7):939-44. doi: 10.1212/wnl.34.7.939. PMID 6610841
- [Background] Mohs RC, Rosen WG, Davis KL. The Alzheimer's disease assessment scale: an instrument for assessing treatment efficacy. Psychopharmacol Bull. 1983;19(3):448-50. No abstract available. PMID 6635122
- [Background] Molloy DW, Standish TI. A guide to the standardized Mini-Mental State Examination. Int Psychogeriatr. 1997;9 Suppl 1:87-94; discussion 143-50. doi: 10.1017/s1041610297004754. PMID 9447431
- [Background] Morris JC. The Clinical Dementia Rating (CDR): current version and scoring rules. Neurology. 1993 Nov;43(11):2412-4. doi: 10.1212/wnl.43.11.2412-a. No abstract available. PMID 8232972
- [Background] Morris JC, Heyman A, Mohs RC, Hughes JP, van Belle G, Fillenbaum G, Mellits ED, Clark C. The Consortium to Establish a Registry for Alzheimer's Disease (CERAD). Part I. Clinical and neuropsychological assessment of Alzheimer's disease. Neurology. 1989 Sep;39(9):1159-65. doi: 10.1212/wnl.39.9.1159. PMID 2771064
- [Background] Ogasawara K, Noda A, Yasuda S, Kobayashi M, Yukawa H, Ogawa A. Effect of calcium antagonist on cerebral blood flow and oxygen metabolism in patients with hypertension and chronic major cerebral artery occlusion: a positron emission tomography study. Nucl Med Commun. 2003 Jan;24(1):71-6. doi: 10.1097/00006231-200301000-00017. PMID 12501022
- [Background] Ohtsuka M, Ono T, Hiroi J, Esumi K, Kikuchi H, Kumada S. Comparison of the cardiovascular effect of FR34235, a new dihydropyridine, with other calcium antagonists. J Cardiovasc Pharmacol. 1983 Nov-Dec;5(6):1074-82. doi: 10.1097/00005344-198311000-00024. PMID 6196557
- [Background] Parry SW, Steen N, Baptist M, Fiaschi KA, Parry O, Kenny RA. Cerebral autoregulation is impaired in cardioinhibitory carotid sinus syndrome. Heart. 2006 Jun;92(6):792-7. doi: 10.1136/hrt.2004.053348. Epub 2006 Jan 31. PMID 16449521
- [Background] Rosenthal J. Nilvadipine: profile of a new calcium antagonist. An overview. J Cardiovasc Pharmacol. 1994;24 Suppl 2:S92-107. PMID 7898101
- [Background] Shimamoto H, Shimamoto Y. Nilvadipine increases cerebral blood flow in elderly hypertensives: comparison with nifedipine. J Hum Hypertens. 1995 Apr;9(4):271-9. PMID 7595910
- [Background] Tollefson GD. Short-term effects of the calcium channel blocker nimodipine (Bay-e-9736) in the management of primary degenerative dementia. Biol Psychiatry. 1990 May 15;27(10):1133-42. doi: 10.1016/0006-3223(90)90050-c. PMID 2187540
- [Background] Verghese J, Lipton RB, Katz MJ, Hall CB, Derby CA, Kuslansky G, Ambrose AF, Sliwinski M, Buschke H. Leisure activities and the risk of dementia in the elderly. N Engl J Med. 2003 Jun 19;348(25):2508-16. doi: 10.1056/NEJMoa022252. PMID 12815136
- [Background] Yasar S, Corrada M, Brookmeyer R, Kawas C. Calcium channel blockers and risk of AD: the Baltimore Longitudinal Study of Aging. Neurobiol Aging. 2005 Feb;26(2):157-63. doi: 10.1016/j.neurobiolaging.2004.03.009. PMID 15582745
- [Derived] Dyer AH, Lawlor B, Kennelly SP; NILVAD Study Group. Gait speed, cognition and falls in people living with mild-to-moderate Alzheimer disease: data from NILVAD. BMC Geriatr. 2020 Mar 30;20(1):117. doi: 10.1186/s12877-020-01531-w. PMID 32228468
- [Derived] Abdullah L, Crawford F, Tsolaki M, Borjesson-Hanson A, Olde Rikkert M, Pasquier F, Wallin A, Kennelly S, Ait-Ghezala G, Paris D, Hendrix S, Blennow K, Lawlor B, Mullan M. The Influence of Baseline Alzheimer's Disease Severity on Cognitive Decline and CSF Biomarkers in the NILVAD Trial. Front Neurol. 2020 Mar 6;11:149. doi: 10.3389/fneur.2020.00149. eCollection 2020. PMID 32210906
- [Derived] de Heus RAA, Olde Rikkert MGM, Tully PJ, Lawlor BA, Claassen JAHR; NILVAD Study Group. Blood Pressure Variability and Progression of Clinical Alzheimer Disease. Hypertension. 2019 Nov;74(5):1172-1180. doi: 10.1161/HYPERTENSIONAHA.119.13664. Epub 2019 Sep 23. PMID 31542965
- [Derived] de Jong DLK, de Heus RAA, Rijpma A, Donders R, Olde Rikkert MGM, Gunther M, Lawlor BA, van Osch MJP, Claassen JAHR. Effects of Nilvadipine on Cerebral Blood Flow in Patients With Alzheimer Disease. Hypertension. 2019 Aug;74(2):413-420. doi: 10.1161/HYPERTENSIONAHA.119.12892. Epub 2019 Jun 17. PMID 31203725
- [Derived] de Heus RAA, Donders R, Santoso AMM, Olde Rikkert MGM, Lawlor BA, Claassen JAHR; Nilvad Study Group. Blood Pressure Lowering With Nilvadipine in Patients With Mild-to-Moderate Alzheimer Disease Does Not Increase the Prevalence of Orthostatic Hypotension. J Am Heart Assoc. 2019 May 21;8(10):e011938. doi: 10.1161/JAHA.119.011938. PMID 31088188
- [Derived] Lawlor B, Segurado R, Kennelly S, Olde Rikkert MGM, Howard R, Pasquier F, Borjesson-Hanson A, Tsolaki M, Lucca U, Molloy DW, Coen R, Riepe MW, Kalman J, Kenny RA, Cregg F, O'Dwyer S, Walsh C, Adams J, Banzi R, Breuilh L, Daly L, Hendrix S, Aisen P, Gaynor S, Sheikhi A, Taekema DG, Verhey FR, Nemni R, Nobili F, Franceschi M, Frisoni G, Zanetti O, Konsta A, Anastasios O, Nenopoulou S, Tsolaki-Tagaraki F, Pakaski M, Dereeper O, de la Sayette V, Senechal O, Lavenu I, Devendeville A, Calais G, Crawford F, Mullan M; NILVAD Study Group. Nilvadipine in mild to moderate Alzheimer disease: A randomised controlled trial. PLoS Med. 2018 Sep 24;15(9):e1002660. doi: 10.1371/journal.pmed.1002660. eCollection 2018 Sep. PMID 30248105